CLINICAL TRIAL: NCT00287248
Title: Evaluation of [123I] IMPY and SPECT as a Marker of Beta-amyloid Protein Deposition in the Brain of Healthy Subjects and Patients With Alzheimer Disease
Brief Title: Assess 123-I IMPY and SPECT Imaging as a Tool to Detect β-Amyloid in the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Alzheimer's Association (Other); Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMYLOID001
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Alzheimer disease; Alzheimer disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Iodine-123; 2,3-dihydro-1H-imidazo(1,2-b)pyrazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [123I] IMPY & SPECT Imaging (Experimental): To assess [123I] IMPY & SPECT Imaging
  Interventions: Drug: [123I] IMPY & SPECT Imaging

INTERVENTIONS:
Drug: [123I] IMPY & SPECT Imaging — Subjects will be injected with 7mCi of [123I]IMPY, followed by SPECT imaging

SUMMARY:
This research is designed to obtain efficacy and safety information for 123-I IMPY as an imaging biomarker for Alzheimer's disease (AD). The distribution of this agent will be measured by obtaining single photon emission computed tomography (SPECT) images of the brain serially over time to determine the relative localization of the radiopharmaceutical in regions of the cortex relative to background regions and develop an optimal technique of radiotracer administration (bolus or bolus with constant infusion). The researchers will then evaluate the utility of 123-I IMPY and SPECT in AD patients as an early diagnostic tool and subsequently serial evaluations of AD patients will be performed to determine if this technique may be useful as a tool for evaluation of progressive brain β-amyloid deposition in AD.

DETAILED DESCRIPTION:
All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImanging (MNI) in New Haven, CT. Approximately 25 patients with mild to moderate Alzheimer's disease (AD) and 20 healthy controls will be recruited to participate in this study. AD patients will be eligible to participate if they have a diagnosis of AD of less than 3 years duration. Healthy controls will be examined to ensure that there is no evidence of neurodegenerative changes including cognitive decline. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be asked to undergo either a bolus injection or bolus injection followed by continuous infusion of 123-I IMPY. Following injection, subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I IMPY in plasma (both protein bound and free) over a 3.5 - 8 hour period. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I IMPY.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRA) criteria.
* Mini-Mental Status Exam score > 16 and < 25.
* Patients have a diagnosis of probable AD for < 3 years prior to screening.

Exclusion Criteria:

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
* Subjects with an iodine allergy.
* The subject has a clinically significant clinical laboratory value and/or medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant thyroid disease, gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other medical or psychiatric disorder.
* The subject has received an investigational drug within 60 days before the screening visit.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Does 123-I IMPY demonstrate qualitatively increased radiotracer uptake in cortical regions consistent with β-amyloid deposition in AD patients relative to controls | 2 years

SECONDARY OUTCOMES:
Can 123-I IMPY and SPECT provide a quantitative and reproducible measure of amyloid deposition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Bacskai BJ, Kajdasz ST, Christie RH, Carter C, Games D, Seubert P, Schenk D, Hyman BT. Imaging of amyloid-beta deposits in brains of living mice permits direct observation of clearance of plaques with immunotherapy. Nat Med. 2001 Mar;7(3):369-72. doi: 10.1038/85525. No abstract available. PMID 11231639
- [Background] Bard F, Barbour R, Cannon C, Carretto R, Fox M, Games D, Guido T, Hoenow K, Hu K, Johnson-Wood K, Khan K, Kholodenko D, Lee C, Lee M, Motter R, Nguyen M, Reed A, Schenk D, Tang P, Vasquez N, Seubert P, Yednock T. Epitope and isotype specificities of antibodies to beta -amyloid peptide for protection against Alzheimer's disease-like neuropathology. Proc Natl Acad Sci U S A. 2003 Feb 18;100(4):2023-8. doi: 10.1073/pnas.0436286100. Epub 2003 Feb 3. PMID 12566568
- [Background] Bard F, Cannon C, Barbour R, Burke RL, Games D, Grajeda H, Guido T, Hu K, Huang J, Johnson-Wood K, Khan K, Kholodenko D, Lee M, Lieberburg I, Motter R, Nguyen M, Soriano F, Vasquez N, Weiss K, Welch B, Seubert P, Schenk D, Yednock T. Peripherally administered antibodies against amyloid beta-peptide enter the central nervous system and reduce pathology in a mouse model of Alzheimer disease. Nat Med. 2000 Aug;6(8):916-9. doi: 10.1038/78682. PMID 10932230
- [Background] Cai L, Chin FT, Pike VW, Toyama H, Liow JS, Zoghbi SS, Modell K, Briard E, Shetty HU, Sinclair K, Donohue S, Tipre D, Kung MP, Dagostin C, Widdowson DA, Green M, Gao W, Herman MM, Ichise M, Innis RB. Synthesis and evaluation of two 18F-labeled 6-iodo-2-(4'-N,N-dimethylamino)phenylimidazo[1,2-a]pyridine derivatives as prospective radioligands for beta-amyloid in Alzheimer's disease. J Med Chem. 2004 Apr 22;47(9):2208-18. doi: 10.1021/jm030477w. PMID 15084119
- [Background] Cummings JL. Alzheimer's disease. N Engl J Med. 2004 Jul 1;351(1):56-67. doi: 10.1056/NEJMra040223. No abstract available. PMID 15229308
- [Background] DeMattos RB, Bales KR, Cummins DJ, Dodart JC, Paul SM, Holtzman DM. Peripheral anti-A beta antibody alters CNS and plasma A beta clearance and decreases brain A beta burden in a mouse model of Alzheimer's disease. Proc Natl Acad Sci U S A. 2001 Jul 17;98(15):8850-5. doi: 10.1073/pnas.151261398. Epub 2001 Jul 3. PMID 11438712
- [Background] DeMattos RB, Bales KR, Cummins DJ, Paul SM, Holtzman DM. Brain to plasma amyloid-beta efflux: a measure of brain amyloid burden in a mouse model of Alzheimer's disease. Science. 2002 Mar 22;295(5563):2264-7. doi: 10.1126/science.1067568. PMID 11910111
- [Background] Dodart JC, Bales KR, Gannon KS, Greene SJ, DeMattos RB, Mathis C, DeLong CA, Wu S, Wu X, Holtzman DM, Paul SM. Immunization reverses memory deficits without reducing brain Abeta burden in Alzheimer's disease model. Nat Neurosci. 2002 May;5(5):452-7. doi: 10.1038/nn842. PMID 11941374
- [Background] Ferrer I, Boada Rovira M, Sanchez Guerra ML, Rey MJ, Costa-Jussa F. Neuropathology and pathogenesis of encephalitis following amyloid-beta immunization in Alzheimer's disease. Brain Pathol. 2004 Jan;14(1):11-20. doi: 10.1111/j.1750-3639.2004.tb00493.x. PMID 14997933
- [Background] Folstein MF, Folstein SE, McHugh PR.
- [Background] Foster DM. Developing and testing integrated multicompartment models to describe a single-input multiple-output study using the SAAM II software system. Adv Exp Med Biol. 1998;445:59-78. doi: 10.1007/978-1-4899-1959-5_4. PMID 9781382
- [Background] Fox NC, Black RS, Gilman S, Rossor MN, Griffith SG, Jenkins L, Koller M; AN1792(QS-21)-201 Study. Effects of Abeta immunization (AN1792) on MRI measures of cerebral volume in Alzheimer disease. Neurology. 2005 May 10;64(9):1563-72. doi: 10.1212/01.WNL.0000159743.08996.99. PMID 15883317
- [Background] Frank RA, Galasko D, Hampel H, Hardy J, de Leon MJ, Mehta PD, Rogers J, Siemers E, Trojanowski JQ; National Institute on Aging Biological Markers Working Group. Biological markers for therapeutic trials in Alzheimer's disease. Proceedings of the biological markers working group; NIA initiative on neuroimaging in Alzheimer's disease. Neurobiol Aging. 2003 Jul-Aug;24(4):521-36. doi: 10.1016/s0197-4580(03)00002-2. No abstract available. PMID 12714109
- [Background] Gilman S, Koller M, Black RS, Jenkins L, Griffith SG, Fox NC, Eisner L, Kirby L, Rovira MB, Forette F, Orgogozo JM; AN1792(QS-21)-201 Study Team. Clinical effects of Abeta immunization (AN1792) in patients with AD in an interrupted trial. Neurology. 2005 May 10;64(9):1553-62. doi: 10.1212/01.WNL.0000159740.16984.3C. PMID 15883316
- [Background] Hardy J, Selkoe DJ. The amyloid hypothesis of Alzheimer's disease: progress and problems on the road to therapeutics. Science. 2002 Jul 19;297(5580):353-6. doi: 10.1126/science.1072994. PMID 12130773
- [Background] Hock C, Konietzko U, Papassotiropoulos A, Wollmer A, Streffer J, von Rotz RC, Davey G, Moritz E, Nitsch RM. Generation of antibodies specific for beta-amyloid by vaccination of patients with Alzheimer disease. Nat Med. 2002 Nov;8(11):1270-5. doi: 10.1038/nm783. Epub 2002 Oct 15. PMID 12379846
- [Background] Hock C, Konietzko U, Streffer JR, Tracy J, Signorell A, Muller-Tillmanns B, Lemke U, Henke K, Moritz E, Garcia E, Wollmer MA, Umbricht D, de Quervain DJ, Hofmann M, Maddalena A, Papassotiropoulos A, Nitsch RM. Antibodies against beta-amyloid slow cognitive decline in Alzheimer's disease. Neuron. 2003 May 22;38(4):547-54. doi: 10.1016/s0896-6273(03)00294-0. PMID 12765607
- [Background] Holtzman DM. Role of apoe/Abeta interactions in the pathogenesis of Alzheimer's disease and cerebral amyloid angiopathy. J Mol Neurosci. 2001 Oct;17(2):147-55. doi: 10.1385/JMN:17:2:147. PMID 11816788
- [Background] Jost BC, Grossberg GT. The natural history of Alzheimer's disease: a brain bank study. J Am Geriatr Soc. 1995 Nov;43(11):1248-55. doi: 10.1111/j.1532-5415.1995.tb07401.x. PMID 7594159
- [Background] Kung HF, Kung MP, Zhuang ZP, Hou C, Lee CW, Plossl K, Zhuang B, Skovronsky DM, Lee VM, Trojanowski JQ. Iodinated tracers for imaging amyloid plaques in the brain. Mol Imaging Biol. 2003 Nov-Dec;5(6):418-26. doi: 10.1016/j.mibio.2003.09.003. PMID 14667496
- [Background] Kung MP, Hou C, Zhuang ZP, Cross AJ, Maier DL, Kung HF. Characterization of IMPY as a potential imaging agent for beta-amyloid plaques in double transgenic PSAPP mice. Eur J Nucl Med Mol Imaging. 2004 Aug;31(8):1136-45. doi: 10.1007/s00259-004-1487-z. Epub 2004 Mar 9. PMID 15007564
- [Background] Kung MP, Hou C, Zhuang ZP, Zhang B, Skovronsky D, Trojanowski JQ, Lee VM, Kung HF. IMPY: an improved thioflavin-T derivative for in vivo labeling of beta-amyloid plaques. Brain Res. 2002 Nov 29;956(2):202-10. doi: 10.1016/s0006-8993(02)03436-4. PMID 12445687
- [Background] Kung MP, Hou C, Zhuang ZP, Skovronsky D, Kung HF. Binding of two potential imaging agents targeting amyloid plaques in postmortem brain tissues of patients with Alzheimer's disease. Brain Res. 2004 Oct 29;1025(1-2):98-105. doi: 10.1016/j.brainres.2004.08.004. PMID 15464749
- [Background] Kung MP, Zhuang ZP, Hou C, Kung HF. Development and evaluation of iodinated tracers targeting amyloid plaques for SPECT imaging. J Mol Neurosci. 2004;24(1):49-53. doi: 10.1385/JMN:24:1:049. PMID 15314249
- [Background] Kung MP, Zhuang ZP, Hou C, Jin LW, Kung HF. Characterization of radioiodinated ligand binding to amyloid beta plaques. J Mol Neurosci. 2003;20(3):249-54. doi: 10.1385/JMN:20:3:249. PMID 14501004
- [Background] Loevinger R, Budinger T, Watson E: MIRD Primer for Absorbed Dose Calculations, Society of Nuclear Medicine, 1988.
- [Background] Masliah E, Hansen L, Adame A, Crews L, Bard F, Lee C, Seubert P, Games D, Kirby L, Schenk D. Abeta vaccination effects on plaque pathology in the absence of encephalitis in Alzheimer disease. Neurology. 2005 Jan 11;64(1):129-31. doi: 10.1212/01.WNL.0000148590.39911.DF. PMID 15642916
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Mohs RC, Knopman D, Petersen RC, Ferris SH, Ernesto C, Grundman M, Sano M, Bieliauskas L, Geldmacher D, Clark C, Thal LJ. Development of cognitive instruments for use in clinical trials of antidementia drugs: additions to the Alzheimer's Disease Assessment Scale that broaden its scope. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S13-21. PMID 9236948
- [Background] Nicoll JA, Wilkinson D, Holmes C, Steart P, Markham H, Weller RO. Neuropathology of human Alzheimer disease after immunization with amyloid-beta peptide: a case report. Nat Med. 2003 Apr;9(4):448-52. doi: 10.1038/nm840. Epub 2003 Mar 17. PMID 12640446
- [Background] Okamura N. [In vivo imaging of amyloid plaques in the brain]. Nihon Ronen Igakkai Zasshi. 2004 Mar;41(2):175-8. doi: 10.3143/geriatrics.41.175. Japanese. PMID 15148750
- [Background] Orgogozo JM, Gilman S, Dartigues JF, Laurent B, Puel M, Kirby LC, Jouanny P, Dubois B, Eisner L, Flitman S, Michel BF, Boada M, Frank A, Hock C. Subacute meningoencephalitis in a subset of patients with AD after Abeta42 immunization. Neurology. 2003 Jul 8;61(1):46-54. doi: 10.1212/01.wnl.0000073623.84147.a8. PMID 12847155
- [Background] Pfeifer M, Boncristiano S, Bondolfi L, Stalder A, Deller T, Staufenbiel M, Mathews PM, Jucker M. Cerebral hemorrhage after passive anti-Abeta immunotherapy. Science. 2002 Nov 15;298(5597):1379. doi: 10.1126/science.1078259. No abstract available. PMID 12434053
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Price DL, Sisodia SS, Borchelt DR. Alzheimer disease--when and why? Nat Genet. 1998 Aug;19(4):314-6. doi: 10.1038/1196. No abstract available. PMID 9697686
- [Background] Racke MM, Boone LI, Hepburn DL, Parsadainian M, Bryan MT, Ness DK, Piroozi KS, Jordan WH, Brown DD, Hoffman WP, Holtzman DM, Bales KR, Gitter BD, May PC, Paul SM, DeMattos RB. Exacerbation of cerebral amyloid angiopathy-associated microhemorrhage in amyloid precursor protein transgenic mice by immunotherapy is dependent on antibody recognition of deposited forms of amyloid beta. J Neurosci. 2005 Jan 19;25(3):629-36. doi: 10.1523/JNEUROSCI.4337-04.2005. PMID 15659599
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Rosen WG, Terry RD, Fuld PA, Katzman R, Peck A. Pathological verification of ischemic score in differentiation of dementias. Ann Neurol. 1980 May;7(5):486-8. doi: 10.1002/ana.410070516. PMID 7396427
- [Background] Schenk DB, Rydel RE, May P, Little S, Panetta J, Lieberburg I, Sinha S. Therapeutic approaches related to amyloid-beta peptide and Alzheimer's disease. J Med Chem. 1995 Oct 13;38(21):4141-54. doi: 10.1021/jm00021a001. No abstract available. PMID 7473539
- [Background] Schenk DB, Seubert P, Lieberburg I, Wallace J. beta-peptide immunization: a possible new treatment for Alzheimer disease. Arch Neurol. 2000 Jul;57(7):934-6. doi: 10.1001/archneur.57.7.934. No abstract available. PMID 10891974
- [Background] Seibyl JP, Zea-Ponce Y, Brenner L, Baldwin RM, Krystal JH, Offord SJ, Mochoviak S, Charney DS, Hoffer PB, Innis RB. Continuous intravenous infusion of iodine-123-IBZM for SPECT determination of human brain dopamine receptor occupancy by antipsychotic agent RWJ-37796. J Nucl Med. 1996 Jan;37(1):11-5. PMID 8543979
- [Background] Seibyl JP, Woods SW, Zoghbi SS, Baldwin RM, Dey HM, Goddard AW, Zea-Ponce Y, Zubal G, Germine M, Smith EO, et al. Dynamic SPECT imaging of dopamine D2 receptors in human subjects with iodine-123-IBZM. J Nucl Med. 1992 Nov;33(11):1964-71. PMID 1432157
- [Background] Stabin MG, Sparks RB, Crowe E. OLINDA/EXM: the second-generation personal computer software for internal dose assessment in nuclear medicine. J Nucl Med. 2005 Jun;46(6):1023-7. PMID 15937315
- [Background] Zhuang ZP, Kung MP, Wilson A, Lee CW, Plossl K, Hou C, Holtzman DM, Kung HF. Structure-activity relationship of imidazo[1,2-a]pyridines as ligands for detecting beta-amyloid plaques in the brain. J Med Chem. 2003 Jan 16;46(2):237-43. doi: 10.1021/jm020351j. PMID 12519062